CLINICAL TRIAL: NCT01192334
Title: Observational Study for Changes of the Single Limb Standing Balance After Total Knee Arthroplasty in Degenerative Osteoarthritis
Brief Title: Changes of the Single Limb Standing Balance After Total Knee Arthroplasty in Degenerative Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Clinical Associate Professor, Ulsan University Hospital
Other Study IDs: chhwang1
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis arthroplasty postural balance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It was well known that total knee arthroplasty could improve the previously impaired proprioception in degenerative osteoarthritis. Most current researches have been focused on the change of the proprioception. However, the evaluation of the proprioception is based on the surrogated end.

Double or single limb standing balance is considered functional scale. It is very important view for the prevention of slipping down injury in evidence-based approaches for knee osteoarthritis.

Unfortunately, few study have been performed for figuring proprioceptive change after surgery out.

Considering the similarity between the proprioception and the standing balance and reported positive result in proprioception after total knee arthroplasty, the investigators supposed that total knee arthroplasty might give an influence on the recovery of single limb standing balance.

ELIGIBILITY:
Inclusion Criteria:

* Medial compartment degenerative knee osteoarthritis showing the varus deformity

Exclusion Criteria:

* History of surgery on the lower extremity except for arthroscopy or menisectomy
* Hip arthritis or, hip or back pain disturbing the standing
* History of participation in sport rehabilitation program within less than 6 months
* Presence of neurological or musculoskeletal disease disturbing the standing
* Patient to reject the participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients to be scheduled to take a elective unilateral total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
single limb standing balance | from issuing admision paper before the surgery up to 4 weeks, average time of this measurement is 2 weeks
  migration distance of center of pressure while single limb standing was recorded through balance performance monitoring
single limb standing balance | from the surgery until the time in which patient shows the same pain score as the pre-operation pain score up to the post-operative 4 weeks, average time of this measurement is post-operative 2 weeks
  migration distance of center of pressure while single limb standing was recorded through balance performance monitoring
single limb standing balance | post-operative 6 months
  migration distance of center of pressure while single limb standing was recorded through balance performance monitoring
single limb standing balance | post-operative 12 months
  migration distance of center of pressure while single limb standing was recorded through balance performance monitoring

SECONDARY OUTCOMES:
balance index | from issuing admision paper before the surgery up to 4 weeks, average time of this measurement is 2 weeks
  balance index, calculated ratio from the deviated distance and time from the neutral point, was collected by using the Biodex machine
balance index | post-operative 6 months
  balance index, calculated ratio from the deviated distance and time from the neutral point, was collected by using the Biodex machine
balance index | post-operative 12 months
  balance index, calculated ratio from the deviated distance and time from the neutral point, was collected by using the Biodex machine

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea